CLINICAL TRIAL: NCT05371938
Title: Longterm Follow up for Displaced Distal Radius Fracture Randomized to Surgery With Volar Locking Plate or External Fixation
Brief Title: Volar Locking Plate Versus External Fixation for Distal Radius Fracture - a Longterm Follow up
Acronym: EXTEND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olof Skoldenberg (Other)
Collaborators: The Swedish Association for Survivors of Accident and Injury (Unknown)
Responsible Party: Sponsor-Investigator, Olof Skoldenberg, Professor, Danderyd Hospital
Organization: Danderyd Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Handledsstudien 1
Record Dates: First submitted 2022-04-01; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Radius Fracture Distal; Surgery; Surgery--Complications; Treatment Complication; Tendon Injuries; Tendon Rupture; Surgical Site Infection; CRPS Type I; CRPS Type II; Dislocation; Osteoarthritis
MeSH Terms: conditions — Wrist Fractures; Tendon Injuries; Surgical Wound Infection; Reflex Sympathetic Dystrophy; Causalgia; Joint Dislocations; Osteoarthritis | interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volar Locking Plate (Experimental): Surgery with volar locking plate
  Interventions: Procedure: Volar locking plate
- External fixation (Active Comparator): Surgery with external fixation
  Interventions: Procedure: external fixation

INTERVENTIONS:
Procedure: Volar locking plate — Volar locking plate is the intervention
  Arms: Volar Locking Plate
Procedure: external fixation — surgery with external fixation
  Arms: External fixation

SUMMARY:
A 10-year follow up of a fusion of two earlier published randomized controlled trials. 203 patients with displaced distal radius fractures were randomized to surgery with a volar locking plate or external fixation.

DETAILED DESCRIPTION:
Follow up includes PROMs (DASH, PRWE, EQ-5D), radiological assesment and objective tests by a hand occupational therapist (ROM, grip strength).

Previous Clinical trials registration for the original studies this long-term follow up is a continuation on: NCT00989222, NCT01034943, NCT01035359

ELIGIBILITY:
Inclusion Criteria:

DS center

* acute unilateral dorsally displaced distal radius fracture with a axial shortening of at least 4 mm or a dorsal displacement of at least 20 degrees.
* Age 20-70

SÖS center

* Age 50-74 for women and 60-74 for men
* injury only after fall from a standing height
* wrist radiography of at least 20 degrees dorsal dislocation and/or at least 5 mm axial shortening
* good knowledge of written and spoken swedish
* fracture diagnosed within 72 hours from injury
* patient resident within the catchment area of SÖS center

Exclusion Criteria:

DS center:

* no previous fracture of either wrist
* ipsilateral acute fracture of the upper extremity
* medicated with warfarin
* unable to cooperate with follow-up (dementia, substance abuse, psychiatric illness, language problems)
* open fracture
* fracture that was not amenable by both methods (distal fragment to small or to comminuted)

SÖS center:

* former disability of either wrist
* other concomitant injuries
* rheumatoid arthritis or other severe joint disorder
* Dementia or pfeiffer score under 5 points
* drug abuse, alcohol abuse or psychiatric disorder
* dependency in activity of daily living
* medical condition contradicting general anesthesia

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Disability of the arm shoulder and hand (DASH) | 10 years after initial surgery
  PROM Patient Rated outcome Measurement. A 30-item questionnaire to assess musculoskeletal disorders in upper limbs. It also has two 4-items optional modules to assess function and symptoms in athletes, artists and workers. Item response range from 1 (no difficult) to 5 (unable). The total score ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
Patient rated wrist evaluation (PRWE) | 10 years after initial surgery
  A patient rated outcome measurement(PROM) a subjective test of function by a 15-item questionnaire. PRWE is specific for wrist evaluation. It consists of two subscales - pain and function. Total score ranges from 0 (no disability) to 100 (severe disability)
Radiological assesment | 10 years after initial surgery
  x-ray of both wrists, AP and lateral. Assessing radial inclination, dorsal tilt, ulnar variance. Osteoarthritis of the radioulnar joint and DRU-joint, fractures in carpus/ulna. VISI/DISI and SL-dissociation.
Objective tests of range of motion (ROM) | 10 years after initial surgery
  pronation and supination, ulnar- and radial deviation, volar flexion and doral extension of both wrists with a goniometer, units will be degrees.
Journal investigation | 0-10 years after initial surgery
  A journal assesment to find complications as infections, reoperations, CRPS, nerv injuries.
EQ-5D | 10 years after initial surgery
  A health related quality of life questionnaire. EQ-5D is the correct name and not an abbreviation. 5 dimensions of health is assessed (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) in three levels (no problems/some or moderate problems/extreme problems). The responses of EQ-5D can be converted to a singel number - a index value and compared with a value set. The index value reflects how good or bad the health statues is. There is also a visual analogue scale on overall health with the scale 0 (worst imaginable health state) to 100 (best imaginable health state).
Objective test of grip strength | 10 year after initial surgery.
  Test of grip strength by GRIPPIT units is Newton. Grip strength will be measured bilateral and presented as maximum, mean and value after 10 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Division of Ortopeadics, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No